CLINICAL TRIAL: NCT07284784
Title: An Open-label Clinical Trial Investigating the Long-term Safety of Buntanetap in Treating Participants With Parkinson's Disease
Brief Title: A Study of Buntanetap in Participants With PD
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Annovis Bio Inc. (Industry)
Collaborators: Duke Clinical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANVS-25002
Record Dates: First submitted 2025-11-26; First posted 2025-12-16 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-11

CONDITIONS: Parkinson's Disease (PD); Deep Brain Stimulation
Keywords: Parkinson's Disease; PD; Deep Brain Stimulation; DBS; buntanetap; Open-Label; posiphen
MeSH Terms: conditions — Parkinson Disease | interventions — phenserine

STUDY DESIGN:
Intervention Model Description: All participants will receive treatment with buntanetap 30 mg daily
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 - buntanetap (Experimental): Cohort 1 will enroll via invitation only for PD participants who have previously participated in bun
  Interventions: Drug: buntanetap/posiphen
- Cohort 2 - buntanetap (Experimental): Cohort 2 will be for PD participants who are receiving deep brain stimulation (DBS) treatment.
  Interventions: Drug: buntanetap/posiphen

INTERVENTIONS:
Drug: buntanetap/posiphen — buntanetap capsules 30 mg by mouth daily

SUMMARY:
This study will examine the long-term safety of buntanetap in participants with PD. This will be a 36-month open-label safety study. This study will be conducted with two cohorts. Cohort 1 will enroll via invitation only for PD participants who have previously participated in buntanetap clinical trials. Cohort 2 will be for PD participants who are receiving deep brain stimulation (DBS) treatment. Qualified participants will receive buntanetap 30mg QD after a screening period of up to 42 days.

DETAILED DESCRIPTION:
This study will examine the long-term safety of buntanetap in participants with PD. This will be a 36-month open-label safety study. This study will be conducted with two cohorts. Cohort 1 will enroll via invitation only for PD participants who have previously participated in buntanetap clinical trials. Cohort 2 will be for PD participants who are receiving deep brain stimulation (DBS) treatment. Qualified participants will receive buntanetap 30mg QD after a screening period of up to 42 days. MMSE, MoCA, C-SSRS, and MDS-UPDRS will be assessed by clinicians who have successfully completed the requisite certifications/trainings for each assessment. Each participant shall be assessed by the same clinician throughout the study. Cohort 1 participants will stop standard of care Parkinson's medications 12h before baseline and annual clinical visits to ensure clinical OFF-state during visit. Cohort 2 participants will stop standard of care Parkinson's medications 12h before all clinic visits. The night before the baseline and annual clinic visits (or early termination visit), Cohort 2 participants will return DBS settings to their initial baseline settings.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of idiopathic PD according to MDS Clinical Diagnostic Criteria for Parkinson's Disease (Postuma et al., 2015) and

   a. Cohort 1: Participated in a prior PD clinical trial with buntanetap. i. A legally authorized representative is required for any participant whose MMSE <21 at screening.

   b. Cohort 2: Has been receiving DBS treatment in either 1) the subthalamic nucleus or 2) the globus pallidus internus for at least 12 months after a successful DBS surgery that achieved the goal.

   i. Female or male adults aged 40 to 85 years. ii. H&Y stage 1-3 in ON state. iii. MMSE 21-30 at screening and baseline.
2. Have a support person who will accompany the participant on study visits at designated times.
3. Female participants of childbearing potential* must have a negative urine pregnancy test at screening, must be non-lactating, and must agree to use a highly effective method of contraception (i.e., a method resulting in a failure rate of less than 1% per year when used consistently and correctly) during the trial and for one month after the last dose of trial treatment, such as:

   1. Oral, intravaginal, or transdermal combined (estrogen plus progestogen) hormonal contraception associated with inhibition of ovulation,
   2. Oral, injectable, or implantable progestogen-only hormonal contraception associated with inhibition of ovulation,
   3. Intrauterine device (IUD),
   4. Intrauterine hormone-releasing system (IUS),
   5. Bilateral tubal occlusion,
   6. Vasectomized partner (a vasectomized partner is a highly effective contraception method provided that the partner is the sole male sexual partner of the participant, and the absence of sperm has been confirmed. If not, an additional highly effective method of contraception should be used),
   7. Sexual abstinence (sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatment. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the study and the preferred and usual lifestyle of the participant).

      * Non-childbearing potential includes surgically sterilized or postmenopausal with no menstrual bleeding for at least one year prior to study start.

   Protocol ANVS-25002 Ver. 2.1; 09-23-2025 Confidential Page 30 of 54
4. Male participants must be sterile or sexually inactive or agree not to father a child during the study and one month after the last dose of study medication and must agree to use a barrier method for contraception. Female partners of male participants must adopt a highly effective method of contraception with a failure rate of less than 1% per year when used consistently and correctly such as:

   1. Oral, intravaginal, or transdermal combined (estrogen plus progestogen) hormonal contraception associated with inhibition of ovulation,
   2. Oral, injectable, or implantable progestogen-only hormonal contraception associated with inhibition of ovulation,
   3. IUD,
   4. IUS,
   5. Bilateral tubal occlusion.
5. No evidence of current suicidal ideation or previous suicide attempt in the past month as evaluated in the C-SSRS.
6. Stability of permitted medications for at least 4 weeks prior to screening. Refer to Concomitant Medications section above for details on prohibited and permitted medications.

   1. Standard of care anti-parkinsonian medication,
   2. Cholinesterase inhibitors and/or memantine medication,
   3. Anticonvulsant medications used for epilepsy or mood stabilization, or neuropathic pain indications, and have not had a breakthrough seizure 3 years prior to screening,
   4. Mood-stabilizing psychotropic agents including, but not limited to, lithium,
7. Adequate visual and hearing ability (physical ability to perform all the study assessments).
8. Good general health with no disease expected to interfere with the study.

Exclusion Criteria:

1. Cohort 1 only: Is currently receiving DBS treatment. (Participant may enroll in Cohort 2 if they meet the corresponding inclusion/exclusion criteria).
2. A history of psychiatric disorder such as schizophrenia, bipolar disorder, or major depression according to the criteria of the most current version of the Diagnostic and Statistical Manual of Mental Disorders (DSM), unless their symptoms have been mild, and they are stable on treatment or no longer need treatment. Mild depression or history of depression that is stable on treatment with selective serotonin reuptake inhibitors (SSRI) or serotonin and norepinephrine reuptake inhibitors (SNRI) medication at a stable dose is acceptable. Refer to Concomitant Medications section above for details on prohibited and permitted medications.
3. A history of seizure disorder. If stable on medication, it is acceptable. Refer to Concomitant Medications section above for details on prohibited and permitted medications.
4. A history or current evidence of long QT syndrome, Fridericia's formula corrected QT (QTcF) interval ≥ 450 ms for men and ≥ 460 ms for women, or torsades de pointes.
5. Bradycardia (<50 bpm) or tachycardia (>100 bpm) on the ECG at screening and deemed medically significant by the PI.

   Protocol ANVS-25002 Ver. 2.1; 09-23-2025 Confidential Page 31 of 54
6. Uncontrolled Type-1 or Type-2 diabetes. A participant with hemoglobin subunit alpha 1c (HbA1c) levels up to 7.5% can be enrolled if the investigator believes the participant's diabetes is under control.
7. Clinically significant renal (Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] <50 mL/min/BSA [body surface area]) or hepatic impairment (Alkaline phosphatase [ALP] > 2.0X the upper limit of normal [ULN] and/or total bilirubin > 2.0X ULN).
8. Any clinically significant abnormal laboratory values. Participants with liver function tests (aspartate aminotransferase [AST] or alanine aminotransferase [ALT]) greater than twice ULN will be excluded.
9. Is at imminent risk of self-harm, based on clinical interview and responses on the C-SSRS, or of harm to others in the opinion of the investigators. Participants must be excluded if they report suicidal ideation with intent, with or without a plan or method (e.g., positive response to Items 4 or 5 in assessment of suicidal ideation on C-SSRS) in the past 2 months, or suicidal behavior in the past 6 months.
10. Cancer or has had a malignant tumor within the past year, except participants who underwent potentially curative therapy with no evidence of recurrence (participants with stable untreated cancer are not excluded).
11. Alcohol / Substance use disorder, moderate to severe, in the last 5 years according to the most current version of the DSM.
12. Participation in another clinical trial with an investigational agent and have taken at least one dose of study medication, unless unblinded on placebo, within 4 weeks prior to the start of screening, or five half-lives of the investigational drug, whichever is greater. The end of a previous investigational trial is the date the last dose of an investigational agent was taken.
13. A learning disability or developmental delay.
14. Participants whom the site PI deems to be otherwise ineligible.
15. A known allergy to the investigational drug or any of its components.

    Inactive ingredients of the investigational medicinal product:
    * Silicified microcrystalline cellulose
    * Dibasic calcium phosphate dihydrate
    * Mannitol
    * Stearic acid
    * Hypromellose (capsule shells structure)
    * Titanium dioxide (opacifier of the capsule shells)
16. Is currently pregnant, breast-feeding, and/or lactating.
17. Uncontrolled hypertension (systolic >160mmHg and/or diastolic >95mmHg) or hypotension (systolic <90mmHg and/or diastolic <60 mmHg) and deemed medically significant by the PI.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2026-01-09 (Actual); Primary Completion 2029-09 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
Safety of buntanetap | 36-months of treatment
  Safety assessments of participants with PD receiving treatment with buntanetap
Adverse Events (AE) | 36-months of treatment
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention
Treatment Emergent Adverse Events (TEAE) | 36-months of treatment
  TEAE is an event that emerges during treatment, having been absent pretreatment, or worsens relative to the pretreatment state
Serious Adverse Events (SAE) | 36-months of treatment
  SAE is defined as any untoward medical occurrence that results in death, is life-threatening, requires inpatient hospitalization, or prolongation of an existing hospitalization, results in persistent or significant disability or incapacity, is a birth defect or congenital anomaly

CONTACTS AND LOCATIONS:
Overall Officials: Laurie Sanders, Ph.D., Principal Investigator — Duke Clinical Research Institute
Locations (25):
- United States (25):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Banner Sun Health Research Institute - Cleo Roberts Center for Clinical Research, Sun City, Arizona
  - Parkinson's & Movement Disorder Institute (PMDI) - Orange County Office, Fountain Valley, California
  - Cenexel Rocky Mountain Clinical Research, Englewood, Colorado
  - First Choice Neurology - Aventura Neurologic Associates, Aventura, Florida
  - Arrow Clinical Trials, Daytona Beach, Florida
  - Accel Clinical Sites-Georgia LLC dba Accel Research Sites-Lake Oconee CRU, DeLand, Florida
  - Renstar Medical Research, Ocala, Florida
  - University of South Florida (USF) - University of South Florida College of Medicine - Parkinson's Di, Tampa, Florida
  - Conquest Research, Winter Park, Florida
  - iResearch Atlanta, Decatur, Georgia
  - Josephson Wallack Munshower Neurology, P.C., Indianapolis, Indiana
  - University of Kansas Medical Center (KUMC) - School of Medicine - Parkinson's Disease and Movement D, Kansas City, Kansas
  - Quest Research Institute, Farmington Hills, Michigan
  - Mount Sinai Hospital, New York, New York
  - Duke Department of Neurosurgery, Durham, North Carolina
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - The Movement Disorder Clinic of Oklahoma, Tulsa, Oklahoma
  - Abington Neurology, Willow Grove, Pennsylvania
  - Medical University of South Carolina (MUSC) - The Murray Center for Research on Parkinson's Disease, Charleston, South Carolina
  - Veracity Neuroscience LLC, Memphis, Tennessee
  - Central Texas Neurology, Round Rock, Texas
  - University of Virginia Health System (UVAHS) - Adult Neurology Clinic, Charlottesville, Virginia
  - Inland Northwest Research, Spokane, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided